CLINICAL TRIAL: NCT03840811
Title: Experimental Human Infection With Isogenic Mutants of Neisseria Gonorrhoeae
Brief Title: Experimental Human Infection With Neisseria Gonorrhoeae
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 09-0106
Record Dates: First submitted 2019-02-07; First posted 2019-02-15 (Actual); Results first posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2020-09-16

CONDITIONS: Gonococcal Infection
Keywords: ceftriaxone; challenge; ciprofloxacin; males; Neisseria gonorrhoeae
MeSH Terms: conditions — Gonorrhea | interventions — Cefixime; Ceftriaxone; Ciprofloxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group 1 (Experimental): Subjects (n = up to 8) will receive a bacterial inoculum containing only the isogenic mutant N. gonorrhoeae strain
  Interventions: Drug: Cefixime; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA7537
- Group 2 (Experimental): Subjects (n = up to 8) will receive a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain.
  Interventions: Drug: Cefixime; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090 A26
- Group 3 (Experimental): Subjects (n= up to 16) will receive a bacterial inoculum containing a mixture of equivalent numbers the isogenic mutant and WT strain
  Interventions: Drug: Cefixime; Drug: Ceftriaxone; Drug: Ciprofloxacin; Biological: Neisseria gonorrhoeae strain FA1090 A26; Biological: Neisseria gonorrhoeae strain FA7537

INTERVENTIONS:
Drug: Cefixime — Mandatory rescue therapy consisting of cefixime 400 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
Drug: Ceftriaxone — Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
Drug: Ciprofloxacin — Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose: if the subject has a positie test of cure 1 week post initial antibiotic treatment
Biological: Neisseria gonorrhoeae strain FA1090 A26 — 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
  Arms: Group 2; Group 3
Biological: Neisseria gonorrhoeae strain FA7537 — 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter
  Arms: Group 1; Group 3

SUMMARY:
This is a Phase 1, interventional, non-randomized, experimental infection model study with healthy adult males adults (N=32) between the ages of 18-36 at study enrollment. The study is designed to test the requirements of predicted N. gonorrhoeae virulence determinants for gonococcal infection in the male urethra. The duration for all participants will be about 3 weeks. Study duration will be approximately about 18 months for implementation and enrollment. The primary objectives of the present study are to: (1) compare infectivity of different isogenic mutants with wild-type (WT) N. gonorrhoeae in noncompetitive infections and to (2) assess relative fitness of the mutant in competitive infections initiated by inocula containing equivalent numbers of both WT and mutant strains for mutants with WT infectivity.

DETAILED DESCRIPTION:
This is a Phase 1, interventional, non-randomized, experimental infection model study with healthy adult males adults (N=32) between the ages of 18-36 at study enrollment. The study is designed to test the requirements of predicted N. gonorrhoeae virulence determinants for gonococcal infection in the male urethra. For each mutant to be investigated under this protocol, groups of subjects will be enrolled first in noncompetitive infection studies: Group 1 (n = up to 8) will receive a bacterial inoculum containing only the isogenic mutant N. gonorrhoeae strain, and Group 2 (n = up to 8) will receive a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain. If primary and secondary outcomes are not different for the isogenic mutant and WT strains, a group of subjects will be enrolled in competitive infection studies: Group 3 (up to 16) will receive a bacterial inoculum containing a mixture of equivalent numbers the isogenic mutant and WT strain. All subjects will be examined daily for symptoms of infection and receive antibiotic treatment at the end of the inpatient portion of the trial. Within 7 days of antibiotic treatment, subjects will return for a follow-up examination. A final follow-up phone interview will be conducted within 2 weeks of antibiotic treatment. The duration for all participants will be about 3 weeks. Study duration will be approximately about 18 months for implementation and enrollment. The primary objectives of the present study are to: (1) compare infectivity of different isogenic mutants with wild-type (WT) N. gonorrhoeae in noncompetitive infections and to (2) assess relative fitness of the mutant in competitive infections initiated by inocula containing equivalent numbers of both WT and mutant strains for mutants with WT infectivity. Note, competitive infections will not be performed if non-competitive infections are substantially different. If this is the case, there will be no analysis for this primary objective. The study secondary objective is to compare the clinical course of infection with mutant and WT N. gonorrhoeae in noncompetitive infections.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy man > / = 18 and < 36 years old
2. Able and willing to be located easily by providing street address and telephone number (land line and/or cell phone number)
3. Willingness to provide written informed consent
4. Able and willing to attend all study visits including 6-day stay in the Clinical Translational Research Center (CTRC) during the trial (with ability to leave the unit during the day) and follow-up visit during the week after treatment
5. Able and willing to abstain from all sexual activity until completion of the study and the follow-up test for gonorrhea is negative
6. Acceptable medical history by screening evaluation
7. No clinically significant abnormalities on physical exam
8. Urinalysis: leukocyte esterase, and White Blood Cell (WBC) values within normal limits (WNL)
9. CH50 WNL
10. Urine negative for chlamydia, gonorrhea, and trichomonas
11. Negative Human Immunodeficiency Virus (HIV), syphilis, and Hepatitis C (HCV) test results
12. Negative Hepatitis B (HBV) core and surface antibodies or results consistent with immunization (negative HBV core antibody/positive HBV surface antibody)
13. Denies history of Sexually Transmitted Infections (STIs) including gonorrhea, chlamydia, syphilis, HIV, HBV, and HCV
14. Denies history of bleeding diathesis
15. Denies history of seizures (due to reports of seizures with ciprofloxacin)
16. Denies history of cancer, except basal cell carcinoma of the skin > 5 years ago
17. Denies history of drug abuse
18. Denies history of genitourinary surgery

Exclusion Criteria:

1. Student or employee under the direct supervision of any of the study investigators
2. Any known immunodeficiencies including complement deficiency, antibody deficiency, chronic granulomatous disease or Human Immunodeficiency Virus (HIV) infection
3. Psychiatric disorders that, in the opinion of the physician, would interfere with the integrity of the data or volunteer safety
4. Unstable depression (defined as receiving either < 3 months of the same medication (and dose) or a decompensating event during the previous 3 months) or depression that, in the opinion of the investigator, will compromise the subject's ability to comply with protocol requirements
5. Heart murmur or heart disease
6. Anatomic abnormality of the urinary tract
7. Any antibiotic treatment in the past 30 days, or azithromycin in the past 60 days
8. Self-reported chemotherapy within the past year
9. Current steroid use, except for topical application
10. Allergy to penicillin, cephalosporins or ciprofloxacin or to lidocaine
11. Treatment with medications in the previous month that are contraindicated with cefixime, ceftriaxone or ciprofloxacin and that cannot be withheld for the single doses given in this study
12. Serum creatinine level < 0.7 or > 1.75 mg/dL and deemed clinically significant by the study physician
13. Serum ALT level < LLN or > 105 U/L and deemed clinically significant by the study physician
14. WBC count < 2.5 or > 15.0 x 10^9/L and deemed clinically significant by the study physician
15. Absolute neutrophil count (ANC) < 1.5 or > 7.5 x 10^9/L and deemed clinically significant by the study physician Exception: For African Americans, ANC values as low as 1.3 x 10^9/L will be allowed (25)
16. Hemoglobin level < 12.0 g/dL or above ULN and deemed clinically significant by the study physician
17. Urinalysis: Qualitative protein level > 1+ or RBC count > 10/hpf

Medications not permitted with cefixime or ceftriaxone:

1. Warfarin
2. Probenecid
3. Aspirin
4. Diuretics such as furosemide
5. Aminoglycoside antibiotics
6. Chloramphenicol

Medications not permitted with ciprofloxacin:

1. Tizanidine
2. Theophylline
3. Warfarin
4. Glyburide
5. Cyclosporine
6. Probenecid
7. Phenytoin
8. Methotrexate
9. Antacids, multivitamins, and other dietary supplements containing magnesium, calcium, aluminum, iron or zinc
10. Caffeine-containing medications
11. Sucralfate or didanosine chewable or buffered tablets

Ages: 18 Years to 36 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2017-04-23 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of North Carolina Health Care - Infectious Diseases, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Waltmann A, Balthazar JT, Begum AA, Hua N, Jerse AE, Shafer WM, Hobbs MM, Duncan JA. Experimental genital tract infection demonstrates Neisseria gonorrhoeae MtrCDE efflux pump is not required for in vivo human infection and identifies gonococcal colonization bottleneck. PLoS Pathog. 2024 Sep 25;20(9):e1012578. doi: 10.1371/journal.ppat.1012578. eCollection 2024 Sep. PMID 39321205
- [Derived] Waltmann A, Balthazar JT, Begum AA, Hua N, Jerse AE, Shafer WM; UNC-Global Clinical Trials Unit/DMID 09-0106 Study Team; Hobbs MM, Duncan JA. Neisseria gonorrhoeae MtrCDE Efflux Pump During In Vivo Experimental Genital Tract Infection in Men and Mice Reveals the Presence of Within-Host Colonization Bottleneck. medRxiv [Preprint]. 2023 Jun 29:2023.06.23.23291824. doi: 10.1101/2023.06.23.23291824. PMID 37425726

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males aged 18-<36 years old, living in central North Carolina, in general good health with no history of sexually transmitted infection (STIs) were enrolled. Participants were enrolled between 23APR2017 and 10NOV2019.
Groups:
- Mutant FA7537: Participants received a bacterial inoculum containing only the isogenic mtrD mutant N. gonorrhoeae strain.
  Cefixime: Mandatory rescue therapy consisting of cefixime 400 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ceftriaxone: Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ciprofloxacin: Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose: if the participant has a positie test of cure 1 week post initial antibiotic treatment.
  Neisseria gonorrhoeae strain FA7537: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
- Wild-type FA1090: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain.
  Cefixime: Mandatory rescue therapy consisting of cefixime 400 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ceftriaxone: Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ciprofloxacin: Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose: if the participant has a positie test of cure 1 week post initial antibiotic treatment.
  Neisseria gonorrhoeae strain FA1090 A26: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
- Mixed FA1090/FA7537: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic MtrD mutant and WT strain.
  Cefixime: Mandatory rescue therapy consisting of cefixime 400 mg orally in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ceftriaxone: Mandatory rescue therapy consisting of ceftriaxone 250 mg intramuscularly in a single dose: on patient request, at the onset of symptoms or on the 5th study day after inoculation.
  Ciprofloxacin: Mandatory antibiotic treatment failure therapy: Ciprofloxacin 500 mg orally in a single dose: if the participant has a positie test of cure 1 week post initial antibiotic treatment.
  Neisseria gonorrhoeae strain FA1090 A26: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
  Neisseria gonorrhoeae strain FA7537: 0.4 mL of a suspension containing 10^5 - 10^6 CFU of Neisseria gonorrhoeae, in phosphate-buffered saline, delivered to the anterior urethra through a No.8 pediatric French catheter.
Period: Overall Study
Arm/Group | Mutant FA7537 | Wild-type FA1090 | Mixed FA1090/FA7537
Started | 9 | 6 | 12
Completed | 9 | 6 | 11
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population includes all enrolled participants.
Groups:
- Mutant FA7537: Participants received a bacterial inoculum containing only the isogenic MtrD mutant N. gonorrhoeae strain.
- Wild-type FA1090: Participants received a bacterial inoculum containing only the wild-type (WT) N. gonorrhoeae strain.
- Mixed FA1090/FA7537: Participants received a bacterial inoculum containing a mixture of equivalent numbers the isogenic MtrD mutant and WT strain.
- Total: Total of all reporting groups
Arm/Group | Mutant FA7537 | Wild-type FA1090 | Mixed FA1090/FA7537 | Total
Number analyzed (Participants) | 9 | 6 | 12 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.2 (6.1) | 21.8 (2.8) | 25.2 (4.7) | 24.4 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 9 | 6 | 12 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 0 | 3
  Not Hispanic or Latino | 7 | 5 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 5 | 5
  White | 6 | 5 | 5 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 12 | 27

OUTCOME MEASURES:

1. Primary Outcome: The Competitive Index of the Mutant Compared to Wild Type Proportion of Organisms With the Predicted Competitive Advantage Recovered From Urine and/or Urethral Swab Specimens From Infected Participants
Description: The competitive index (CI) is defined by the ratio of colony forming units (cfu) of the two strains recovered from urine cultures on the day of treatment (output) compared to the ratio of strains in the inoculum (input):
  CI = mutant cfu(output)/wild-type cfu(output) ÷ mutant cfu(input)/wild-type cfu(input).
  The CI is used to assess whether the fitness of a given mutant is different than that of wild-type, and CI as a ratio is compared to 1. If it's not significantly different than 1, then no significant difference in the fitness was observed. Mutant or wild-type cfu values of 0 were replaced by 1 in the calculation of competitive index.
  The assessment was performed in the MtrD trial mixed group.
Time Frame: Baseline and the day of treatment, any day between Day 2 and Day 6
Population: The evaluable population included participants who received a dose of N. gonorrhoeae within 1 log10 of the intended dose, reached an objective study endpoint (urethral discharge or day 6), and had a valid competitive index (the competitive index could not be calculated for participant who had a negative urine culture result on the day of treatment).
Measure: Median (Full Range); unit: ratio
Arm/Group | Mixed FA1090/FA7537
Number analyzed (Participants) | 10
ratio | 15.11 [0.01 to 78.93]
Statistical Analysis 1: Comparison: Mixed FA1090/FA7537; To assess whether the fitness of a given mutant is different than that of wild-type, the ratio of colony-forming units of the mutant strain was compared to those of the WT strain at the time of treatment and in the inoculum using a Wilcoxon Signed-Rank Test with a significance level of 0.025. CIs of participants in Mixed FA1090 + FA7537 group were compared to mean = 1; Test type: Other; p = 0.230, Sign test

2. Primary Outcome: Proportion of Participants That Become Infected as Defined by a Positive Urine or Urethral Swab Culture Among Infections Initiated With Individual N. Gonorrhoeae Strains in Non-competitive Infections
Description: Infection is defined by a positive urine or urethral swab culture. The proportion of infected participants by Day 6 with N. gonorrhoeae was assessed in each trial by group among participants with non-competitive infections. Participants could become infected and received treatment any day before or on day 6.
Time Frame: day of infection, any day between Day 2 and Day 6
Population: The evaluable population included participants who received a dose of N. gonorrhoeae within 1 log10 of the intended dose and reached an objective study endpoint (urethral discharge or day 6).
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mutant FA7537 | Wild-type FA1090
Number analyzed (Participants) | 7 | 6
proportion of participants | 0.86 [0.42 to 1.00] | 1.00 [0.54 to 1.00]
Statistical Analysis 1: Comparison: Mutant FA7537 vs Wild-type FA1090; Test type: Other; p = 0.54, Fisher Exact — One-sided Fisher's Exact Test with alpha=0.025; Risk Difference (RD) = -0.14, 95% CI 2-sided [-0.58 to 0.34]

3. Primary Outcome: Proportion of Participants That Become Infected as Defined by a Positive Urine or Urethral Swab Culture for Infections Initiated With Mixed Inocula
Description: Infection is defined by a positive urine or urethral swab culture. The proportion of infected participants by Day 6 with N. gonorrhoeae was assessed in each trial among participants with infections initiated with mixed inocula. Participants could become infected and received treatment any day before or on day 6.
Time Frame: day of infection, any day between Day 2 and Day 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mixed FA1090/FA7537
Number analyzed (Participants) | 11
proportion of participants | 1.00 [0.72 to 1.00]

4. Secondary Outcome: Median Time From Inoculation to Treatment Among Infected Participants by Day 6, by Strain, in Non-competitive Infections
Description: The median time from inoculation to antibiotic treatment were calculated for each group.
Time Frame: Day 2 through the day of treatment, up to Day 6
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Mutant FA7537 | Wild-type FA1090
Number analyzed (Participants) | 7 | 6
days | 3.0 [1 to 5] | 3.0 [1 to 4]

5. Secondary Outcome: Proportion of Participants With Occurrence of Bacteriuria in Non-competitive Infections, by Strain
Description: Bacteriuria is defined as Log10 cfu N. gonorrhoeae/mL urine sediment.
Time Frame: Day of occurrence, any day between Day 2 and Day 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mutant FA7537 | Wild-type FA1090
Number analyzed (Participants) | 7 | 6
proportion of participants | 0.86 [0.42 to 1.00] | 1.00 [0.54 to 1.00]

6. Secondary Outcome: Proportion of Participants With Occurrence of Signs and Symptoms of Urethritis Attributable to Gonococcal Infection in Non-competitive Infections, by Strain
Description: Participants with any subjective symptoms or objective signs (observed urethral discharge) during period 01 (post-inoculation and before treatment which can occur on or before day 6) from the Solicited Events Form were captured.
Time Frame: Day of occurrence, any day between Day 2 and Day 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mutant FA7537 | Wild-type FA1090
Number analyzed (Participants) | 7 | 6
proportion of participants | 1.00 [0.59 to 1.00] | 1.00 [0.54 to 1.00]

7. Secondary Outcome: Proportion of Participants With Occurrence of Urethritis in Non-competitive Infections
Description: Urethritis is defined as >= 5.8 Log10 WBC/mL urine sediment.
Time Frame: Day of occurrence, any day between Day 2 and Day 6
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Mutant FA7537 | Wild-type FA1090
Number analyzed (Participants) | 7 | 6
proportion of participants | 1.00 [0.59 to 1.00] | 1.00 [0.54 to 1.00]

ADVERSE EVENTS:
Time Frame: All adverse events that occurred from inoculation (Day 1) through the 2 week final follow-up phone call (Study Days 12-23) were reported.
Description: The solicited and unsolicited AEs reported for the MtrD trial were summarized using MedDRA 22.1
Arm/Group | Mutant FA7537 | Wild-type FA1090 | Mixed FA1090/FA7537
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/6 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/12
Other Adverse Events (participants affected / at risk) | 9/9 | 6/6 | 12/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mutant FA7537 (N=9) | Wild-type FA1090 (N=6) | Mixed FA1090/FA7537 (N=12)
Tingling (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Irritation or Itching (Reproductive system and breast disorders) | 2 (2) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 6 (6) | 3 (3) | 6 (6)
Urethral Discharge (Renal and urinary disorders) | 6 (6) | 6 (6) | 12 (13)
Feverishness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Testicular Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2)
Urinary Frequency (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 3 (3) | 3 (3) | 1 (1)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0)
Heart Rate Irregular (Investigations) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Seasonal Allergy (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Urethral Discharge (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urethritis Noninfective (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT03840811/Prot_SAP_000.pdf